CLINICAL TRIAL: NCT04188938
Title: Occult Pneumothorax in Patients With Blunt or Penetrating Trauma: A Descriptive, Cross-sectional Study
Brief Title: Occult Pneumothorax in Patients With Blunt or Penetrating Trauma
Status: Completed | Type: Observational
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Semra Aslay, Ass. Prof. (M.D.), European University of Lefke
Other Study IDs: Pneumothorax
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Pneumothorax; Acute; Trauma Chest
Keywords: Trauma; Thorax; Emergency; Pneumothorax
MeSH Terms: conditions — Pneumothorax; Thoracic Injuries; Wounds and Injuries; Emergencies | interventions — Pneumothorax, Artificial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Occult pneumothorax in trauma patients: Age>16, multi-trauma, consulted thoracic surgeon, underwent CXR- CT.
  Interventions: Other: Evaluation of occult pneumothorax in who had a blunt or penetrating chest trauma

INTERVENTIONS:
Other: Evaluation of occult pneumothorax in who had a blunt or penetrating chest trauma
  Other Names: Trauma; Pneumothorax

SUMMARY:
Pneumothorax is a common life-threatening complication, frequently seen in patients who have been admitted to the emergency department and intensive care unit. This study aimed to describe the features of patients with pneumothorax due to blunt or penetrating trauma. A total of 615 patients admitted to the emergency department between January 2008 and December 2010 due to multi-trauma, and underwent both chest x-ray and computed chest tomography were included in the study. There were 157 patients with a diagnosis of pneumothorax. Fifty-five of them were excluded because of the eligible criteria. The final study population included 105 patients. The computed chest tomography reading was considered as the gold standard for the occult pneumothorax diagnosis. Data on patient characteristics, trauma types, accompanied traumas, etiology of the chest trauma, and chest x-ray, and computed chest tomography results were recorded.

DETAILED DESCRIPTION:
Thoracic injuries are the third most common cause of trauma-related morbidity/mortality and hospitalization after heart disease and malignancies. At least 25% of blunt traumatic deaths are a direct consequence of chest trauma. Additionally, rib fracture and pneumothorax are the first two most frequent blunt thoracic traumas, respectively.

Pneumothorax (PTX) is a common life-threatening complication and frequently seen in patients who have been admitted to the Emergency Department (ED) and Intense Care Units (ICU). Some traumatic PTXs are clinically and radiologically silent, not identified during the initial assessment and cannot be visible on supine chest x-ray (CXR), but later diagnosed by computed tomography (CT). This type of PTX is called occult pneumothorax (OPTX) and has been found in 30-55% of chest trauma cases. The clinical diagnosis of PTX is incorrect in approximately 30% of all traumatic cases. Besides, it has been stated that PTX has the potential to elevate the mortality rate in patients with trauma if it is not quickly managed.

On the other hand, small or medium undetected PTX usually is not life-threatening. However, delays in the diagnosis and management may result in a rapid progression of OPTX to tension PTX and lead to severe dyspnea and even death. Therefore, early detection is crucial and may influence the evaluation and management of PTX and probably be a lifesaving action.

The initial diagnostic screening test of PTX is usually CXR. However, studies reported that CXR is an insensitive and unreliable test. When the chest x-ray of the patient is acquired in a supine position, even if all of the symptoms related to pneumothorax are present (since the air is not located at the apical pulmonary region), there may not be an image consistent with PTX. For this reason, although CXR is usually used for many thoracic injuries as a screening test, it may miss the diagnosis of some thoracic injuries, including rib fractures, pulmonary contusions, and OPTX.

On the other hand, the role of CT in the assessment of chest injuries has expanded considerably in the management of both blunt and penetrating traumas. The increasing use of CT in the evaluation and management of patients with chest trauma has led to correct and sensitive identification of undetected injuries, including OPTX.

There are limited, but conflicting data about the ideal management type of OPTX in blunt trauma. Some physicians prefer the insertion of a tube thoracostomy (TT) for all OPTX patients, while others favor close observation without chest drainage. Physicians who prefer to insert a TT claim that an untreated OPTX can rapidly evolve into a tension PTX with catastrophic consequences. However, those who favor close observation without TT claim that patients should not be subjected to unnecessary invasive processes.

This study aimed to identify the incidence of OPTX in patients with blunt or penetrating trauma.

This study is a single-center (Emergency Department of Ankara Training and Research Hospital) retrospective analysis of trauma registry data. All consecutive participants over the age of 16 who were admitted to the ED between the 1st of January 2008 and 31st of December 2010 due to multi-trauma, consulted by a thoracic surgeon and underwent both CXR and CT were included in the study. Files of 615 patients who were admitted to ED with a thoracic trauma were reviewed (2008; n=187, 2009; n=168, and 2010; n=260). Patients who had no simultaneous CXR+CT or no pathology in their CT were excluded (n=458). Also, patients not referred to a chest surgeon, and those referred to some other hospital were excluded (n=52). Data for the remaining 105 patients were analyzed. The CT interpretation was considered as the gold standard for the PTX diagnosis. Electronic medical records were then searched for patient characteristics (age and gender), trauma types (blunt or penetrating), accompanied traumas (intra-cerebral and intra-abdominal systems), etiology of the chest trauma (traffic accidents, falls, other), and CXR and CT results. Additionally, the intervention types (thoracostomy tube insertion, thoracentesis, no intervention) during the early phase of the management were recorded. All chest x-rays were performed on the supine position based on the trauma protocol of the hospital. Cases missed by the CXR but identified in the CT were defined as OPTX. Using the web-based Java applet developed by Russ Lenth (https://homepage.divms.uiowa.edu/~rlenth/Power/), a post hoc sample size calculation was performed based on a 7% expected prevalence of OPTX. Given an infinite population and a margin of error of 5%, a sample size of 100 cases is required to estimate OPTX in the study population with a confidence interval of 95%. Statistical analysis was performed with the Statistical Package for the Social Sciences version 22 (SPSS, IBM, Armonk, NY, USA). The 'number (n),' 'percentage (%),' 'mean,' and 'standard deviation (SD)' was given for the descriptive statistics. Pearson Chi-Square or Fisher's exact tests used to compare categorical data. Age between groups was analyzed using the Mann-Whitney U test. Logistic regression analysis was applied to check for independent factors affecting the presence of OPTX. The results were evaluated with a confidence interval of 95%, and the level of significance, p, was set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

>16 years of age consulted by a thoracic surgeon had a multi-trauma underwent both chest x ray and computed tomography

Exclusion Criteria:

<16 years of age not consulted by a thoracic surgeon did not have a multi-trauma did not undergo both chest x ray and computed tomography

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive participants over the age of 16 who were admitted to the ED between the 1st of January 2008 and 31st of December 2010 due to multi-trauma, consulted by a thoracic surgeon and underwent both CXR and CT were included in the study.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2011-04-19 (Actual)

PRIMARY OUTCOMES:
Occult Pneumothorax in Patients with Blunt or Penetrating Thoracic Trauma | Through study completion, an average of 1 year
  Patient Registry

CONTACTS AND LOCATIONS:
Overall Officials: Semra Aslay, M.D., Study Director — European University of Lefke

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participating data
Supporting Information: SAP
Time Frame: After published there is no ending time frame
Access Criteria: All consecutive participants over the age of 16 who were admitted to the ED between the 1st of January 2008 and 31st of December 2010 due to multi-trauma, consulted by a thoracic surgeon and underwent both CXR and CT were included in the study.

REFERENCES:
- [Result] Wilson H, Ellsmere J, Tallon J, Kirkpatrick A. Occult pneumothorax in the blunt trauma patient: tube thoracostomy or observation? Injury. 2009 Sep;40(9):928-31. doi: 10.1016/j.injury.2009.04.005. Epub 2009 Jun 17. PMID 19539280
- [Result] Soldati G, Testa A, Sher S, Pignataro G, La Sala M, Silveri NG. Occult traumatic pneumothorax: diagnostic accuracy of lung ultrasonography in the emergency department. Chest. 2008 Jan;133(1):204-11. doi: 10.1378/chest.07-1595. Epub 2007 Oct 9. PMID 17925411
- [Result] Kunitake RC, Kornblith LZ, Cohen MJ, Callcut RA. Trauma Early Mortality Prediction Tool (TEMPT) for assessing 28-day mortality. Trauma Surg Acute Care Open. 2018 Jan 8;3(1):e000131. doi: 10.1136/tsaco-2017-000131. eCollection 2018. PMID 29766125
- [Result] Ding W, Shen Y, Yang J, He X, Zhang M. Diagnosis of pneumothorax by radiography and ultrasonography: a meta-analysis. Chest. 2011 Oct;140(4):859-866. doi: 10.1378/chest.10-2946. Epub 2011 May 5. PMID 21546439
- [Result] Ball CG, Kirkpatrick AW, Laupland KB, Fox DL, Litvinchuk S, Dyer DM, Anderson IB, Hameed SM, Kortbeek JB, Mulloy R. Factors related to the failure of radiographic recognition of occult posttraumatic pneumothoraces. Am J Surg. 2005 May;189(5):541-6; discussion 546. doi: 10.1016/j.amjsurg.2005.01.018. PMID 15862493
- [Result] Chan YH, Zeng YZ, Wu HC, Wu MC, Sun HM. Effective Pneumothorax Detection for Chest X-Ray Images Using Local Binary Pattern and Support Vector Machine. J Healthc Eng. 2018 Apr 3;2018:2908517. doi: 10.1155/2018/2908517. eCollection 2018. PMID 29849996
- [Result] Holmes JF, Brant WE, Bogren HG, London KL, Kuppermann N. Prevalence and importance of pneumothoraces visualized on abdominal computed tomographic scan in children with blunt trauma. J Trauma. 2001 Mar;50(3):516-20. doi: 10.1097/00005373-200103000-00017. PMID 11265032
- [Result] Lee LK, Rogers AJ, Ehrlich PF, Kwok M, Sokolove PE, Blumberg S, Kooistra J, Olsen CS, Wootton-Gorges S, Cooper A, Kuppermann N, Holmes JF; Pediatric Emergency Care Applied Research Network (PECARN). Occult pneumothoraces in children with blunt torso trauma. Acad Emerg Med. 2014 Apr;21(4):440-8. doi: 10.1111/acem.12344. PMID 24730407
- [Result] Akoglu H, Akoglu EU, Evman S, Akoglu T, Denizbasi A, Guneysel O, Onur O, Onur E. Utility of cervical spinal and abdominal computed tomography in diagnosing occult pneumothorax in patients with blunt trauma: Computed tomographic imaging protocol matters. J Trauma Acute Care Surg. 2012 Oct;73(4):874-9. doi: 10.1097/TA.0b013e3182569ff2. PMID 22835995
- [Result] Plurad D, Green D, Demetriades D, Rhee P. The increasing use of chest computed tomography for trauma: is it being overutilized? J Trauma. 2007 Mar;62(3):631-5. doi: 10.1097/TA.0b013e31802bf009. PMID 17414339
- [Result] Enderson BL, Abdalla R, Frame SB, Casey MT, Gould H, Maull KI. Tube thoracostomy for occult pneumothorax: a prospective randomized study of its use. J Trauma. 1993 Nov;35(5):726-9; discussion 729-30. PMID 8230337
- [Result] Ouellet JF, Trottier V, Kmet L, Rizoli S, Laupland K, Ball CG, Sirois M, Kirkpatrick AW. The OPTICC trial: a multi-institutional study of occult pneumothoraces in critical care. Am J Surg. 2009 May;197(5):581-6. doi: 10.1016/j.amjsurg.2008.12.007. PMID 19306978
- [Result] Ball CG, Kirkpatrick AW, Feliciano DV. The occult pneumothorax: what have we learned? Can J Surg. 2009 Oct;52(5):E173-9. PMID 19865549
- [Result] Matsumoto S, Kishikawa M, Hayakawa K, Narumi A, Matsunami K, Kitano M. A method to detect occult pneumothorax with chest radiography. Ann Emerg Med. 2011 Apr;57(4):378-81. doi: 10.1016/j.annemergmed.2010.08.012. Epub 2010 Sep 22. PMID 20864214
- [Result] Ball CG, Kirkpatrick AW, Fox DL, Laupland KB, Louis LJ, Andrews GD, Dunlop MP, Kortbeek JB, Nicolaou S. Are occult pneumothoraces truly occult or simply missed? J Trauma. 2006 Feb;60(2):294-8 discussion 298-9. doi: 10.1097/01.ta.0000202462.96207.18. PMID 16508485
- [Result] Guerrero-Lopez F, Vazquez-Mata G, Alcazar-Romero PP, Fernandez-Mondejar E, Aguayo-Hoyos E, Linde-Valverde CM. Evaluation of the utility of computed tomography in the initial assessment of the critical care patient with chest trauma. Crit Care Med. 2000 May;28(5):1370-5. doi: 10.1097/00003246-200005000-00018. PMID 10834680
- [Result] Kirkpatrick AW, Sirois M, Laupland KB, Liu D, Rowan K, Ball CG, Hameed SM, Brown R, Simons R, Dulchavsky SA, Hamiilton DR, Nicolaou S. Hand-held thoracic sonography for detecting post-traumatic pneumothoraces: the Extended Focused Assessment with Sonography for Trauma (EFAST). J Trauma. 2004 Aug;57(2):288-95. doi: 10.1097/01.ta.0000133565.88871.e4. PMID 15345974
- [Result] Matsumoto S, Sekine K, Funabiki T, Orita T, Shimizu M, Hayashida K, Kazamaki T, Suzuki T, Kishikawa M, Yamazaki M, Kitano M. Diagnostic accuracy of oblique chest radiograph for occult pneumothorax: comparison with ultrasonography. World J Emerg Surg. 2016 Jan 13;11:5. doi: 10.1186/s13017-016-0061-x. eCollection 2016. PMID 26766962
- [Result] Neff MA, Monk JS Jr, Peters K, Nikhilesh A. Detection of occult pneumothoraces on abdominal computed tomographic scans in trauma patients. J Trauma. 2000 Aug;49(2):281-5. doi: 10.1097/00005373-200008000-00015. PMID 10963540
- [Result] Rowan KR, Kirkpatrick AW, Liu D, Forkheim KE, Mayo JR, Nicolaou S. Traumatic pneumothorax detection with thoracic US: correlation with chest radiography and CT--initial experience. Radiology. 2002 Oct;225(1):210-4. doi: 10.1148/radiol.2251011102. PMID 12355007
- [Result] Misthos P, Kakaris S, Sepsas E, Athanassiadi K, Skottis I. A prospective analysis of occult pneumothorax, delayed pneumothorax and delayed hemothorax after minor blunt thoracic trauma. Eur J Cardiothorac Surg. 2004 May;25(5):859-64. doi: 10.1016/j.ejcts.2004.01.044. PMID 15082295
- [Result] Moore FO, Goslar PW, Coimbra R, Velmahos G, Brown CV, Coopwood TB Jr, Lottenberg L, Phelan HA, Bruns BR, Sherck JP, Norwood SH, Barnes SL, Matthews MR, Hoff WS, de Moya MA, Bansal V, Hu CK, Karmy-Jones RC, Vinces F, Pembaur K, Notrica DM, Haan JM. Blunt traumatic occult pneumothorax: is observation safe?--results of a prospective, AAST multicenter study. J Trauma. 2011 May;70(5):1019-23; discussion 1023-5. doi: 10.1097/TA.0b013e318213f727. PMID 21610419
- [Result] Patel BH, Lew CO, Dall T, Anderson CL, Rodriguez R, Langdorf MI. Chest tube output, duration, and length of stay are similar for pneumothorax and hemothorax seen only on computed tomography vs. chest radiograph. Eur J Trauma Emerg Surg. 2021 Aug;47(4):939-947. doi: 10.1007/s00068-019-01198-y. Epub 2019 Aug 5. PMID 31384999
- [Result] Tam MM. Occult pneumothorax in trauma patients: should this be sought in the focused assessment with sonography for trauma examination? Emerg Med Australas. 2005 Oct-Dec;17(5-6):488-93. doi: 10.1111/j.1742-6723.2005.00781.x. PMID 16302942
- [Result] Barry R, Thompson E. Outcomes after rib fractures in geriatric blunt trauma patients. Am J Surg. 2018 Jun;215(6):1020-1023. doi: 10.1016/j.amjsurg.2018.03.011. Epub 2018 Mar 9. PMID 29548528
- [Result] Yang S, Netterwald J, Wang W, Zhu H. Characterization of the elements and proteins responsible for interferon-stimulated gene induction by human cytomegalovirus. J Virol. 2005 Apr;79(8):5027-34. doi: 10.1128/JVI.79.8.5027-5034.2005. PMID 15795288
- [Result] Adolfsson E, Wesolowska P, Izewska J, Lund E, Tedgren AC. END-TO-END AUDIT: COMPARISON OF TLD AND LITHIUM FORMATE EPR DOSIMETRY. Radiat Prot Dosimetry. 2019 Dec 31;186(1):119-122. doi: 10.1093/rpd/ncy289. PMID 30929009